CLINICAL TRIAL: NCT05206396
Title: Do Tumor-Infiltrating Lymphocytes Predict Complete Pathologic Response to Neoadjuvant Systemic Therapy in Breast Cancer Patients?
Brief Title: TIL Relation to pCR After Neoadjuvant Therapy in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Aly, Professor, Ain Shams University
Other Study IDs: R148/2021
Record Dates: First submitted 2022-01-21; First posted 2022-01-25 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: Tumor-infiltrating lymphocytes
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — pre-existing histopathologic samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TIL in breast cancer patients who completed neoadjuvant therapy: * Tumour infiltrating lymphocytes will be examined on pre-existing histopathologic samples.
  * Data will be extracted from the files of the patients including:
  * Demographic data, clinicopathologic data, pathologic complete response, and date of last follow up.
  Interventions: Diagnostic Test: TIL assessment in pre-existing histopathological specimens

INTERVENTIONS:
Diagnostic Test: TIL assessment in pre-existing histopathological specimens — TIL assessment in pre-existing histopathological specimens and their relation to complete pathological response and 1-year invasive disease-free interval

SUMMARY:
Neoadjuvant systemic treatment for breast cancer (used in locally advanced and operable breast cancer) includes anthracycline based chemotherapy (Doxorubicin/Cyclophosphamide) followed by taxanes (weekly Paclitaxel or Docetaxel) with antiHer-2 Trastuzumab or dual antiHer-2 Trastuzumab plus Pertuzumab. Other regimens include Docetaxel plus Carboplatin plus Trastuzumab alone or combined with pertuzumab for Her-2 positive patients.

The tumor microenvironment, which includes extracellular matrix and stromal cells, is a key factor in tumorigenicity and the prediction of the efficacy of immunotherapy, conventional chemotherapy, and other anticancer therapies. Tumor-infiltrating lymphocytes (TILs), one of the most important components of the tumor microenvironment, were reported to predict the response to NAC both for tumors and axillary lymph nodes in breast cancer patients. This study is conducted to examine the relationship between tumor-infiltrating lymphocytes (categorized into three levels) and the pathologic complete response to neoadjuvant systemic therapy in breast cancer patients, and to examine the relationship between TILs and 1-year invasive disease-free survival (IDFS).

DETAILED DESCRIPTION:
Neoadjuvant systemic treatment for breast cancer is used in locally advanced and operable breast cancer. Standard neoadjuvant systemic therapy regimens for breast cancer patients include anthracycline based chemotherapy (Doxorubicin/Cyclophosphamide) followed by taxanes (weekly Paclitaxel or Docetaxel) with antiHer-2 Trastuzumab or dual antiHer-2 Trastuzumab plus Pertuzumab. Other regimens include Docetaxel plus Carboplatin plus Trastuzumab alone or combined with pertuzumab for Her-2 positive patients.

The tumor microenvironment, which includes extracellular matrix and stromal cells, is a key factor in tumorigenicity and the prediction of the efficacy of immunotherapy, conventional chemotherapy, and other anticancer therapies. Tumor-infiltrating lymphocytes (TILs), one of the most important components of the tumor microenvironment, were reported to predict the response to NAC both for tumors and axillary lymph nodes in breast cancer patients. This study is conducted to examine the relationship between tumor-infiltrating lymphocytes (categorized into three levels) and the pathologic complete response to neoadjuvant systemic therapy in breast cancer patients, and to examine the relationship between TILs and 1-year invasive disease-free survival (IDFS).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or more
* Histologically proven invasive breast cancer
* All patients diagnosed with breast cancer except T1N0 and Metastatic breast cancer
* Patients who completed their systemic neoadjuvant therapy

Exclusion Criteria:

* Second malignancy
* Patients who started but didn't complete neoadjuvant systemic therapy
* Patients who didn't undergo surgery after neoadjuvant systemic therapy
* Pregnant patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years old or more, diagnosed with breast cancer fulfilling the inclusion criteria with available histopathological sample and complete medical records will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2022-07-24 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of TIL relation to pathologic complete response | 1 year
  TIL examined from pre-existing histopathological specimens and data of pathologic complete response will be collected from medical records

SECONDARY OUTCOMES:
1-year disease-free interval | 1 year
  1-year disease-free interval will be collected from data in medical records

CONTACTS AND LOCATIONS:
Overall Officials: Iman Sharawy, MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The results of the study will be shared